CLINICAL TRIAL: NCT02965664
Title: A Phase 2a, Double-Masked, Randomized, Placebo-Controlled, Single-Administration Study to Establish Safety, Tolerability and Efficacy of PresbiDrops (CSF-1) in Presbyopic Subjects
Brief Title: Safety, Tolerability and Efficacy of PresbiDrops (CSF-1) in Presbyopic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orasis Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FG-PRE-102
Record Dates: First submitted 2016-11-14; First posted 2016-11-17 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PresbiDrops (CSF-1) (Experimental): Participants self-administer PresbiDrops (CSF-1) , with the supervision or help of the hospital staff - one drop in each eye on the day of treatment
  Interventions: Drug: PresbiDrops (CSF-1)
- Placebo (Placebo Comparator): Participants self-administer Placebo, with the supervision or help of the hospital staff - one drop in each eye on the day of treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PresbiDrops (CSF-1) — PresbiDrops (CSF-1) is a topical ophthalmic drug.
  Arms: PresbiDrops (CSF-1)
Drug: Placebo — Placebo drops contain the same ingredients as PresbiDrops except for the active ingredients
  Arms: Placebo

SUMMARY:
A study to Establish Safety, Tolerability, and Efficacy of PresbiDrops (CSF-1) in Presbyopic Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 40 and 65 years of age (inclusive)
2. Subjects who provide written informed consent to participate in the study
3. Subjects have signs of presbyopia upon ophthalmic examination
4. Subjects have normal presbyopia with no distance correction or with distance refraction, which is within those limits: sphere between +3 Dioptres and -3 Dioptres, cylinder no greater than ± 0.75 DC (based on subjective refraction test)
5. Subjects must have best corrected vision of at least 20/20 in both eyes, and currently depend on reading glasses or bifocals in which the near addition is > +1.00 Dioptres
6. Subjects in general good health in the opinion of the Investigator as determined by medical history
7. Women with childbearing potential must have a negative urine pregnancy test at Screening and be willing and able to use a medically acceptable method of birth control or postmenopausal. Acceptable methods of birth control in this study include: vasectomy, tubal ligation, consistent use of an approved oral contraceptive (birth control pill), intrauterine device, hormonal implants, contraceptive injection or a double barrier method (diaphragm with spermicidal gel or condom with contraceptive foam).

   Postmenopausal women are defined as women with menstruation cessation for 12 consecutive months prior to signing of the informed consent form.
8. Subjects must be able to understand the requirements of the study and must be willing to comply with the requirements of the study

Exclusion Criteria:

1. History of macular disease or any other ocular conditions or congenital malformation
2. Any medical condition known to affect the structure of uvea, cornea, lens or retina or main function of the eyes
3. No cataract or minimal nuclear sclerosis
4. Severe dry eye
5. Any topical ophthalmic medications, other than artificial tears (up to a maximum of 4 times per day) and medications that are associated with fluctuation of accommodative capacity and/or pupil size, unless on a stable dose for at least 3 months before Screening
6. Contact lenses for the past three months before the Screening visit
7. A difference of more than 0.50 Dioptres between the manifest spherical equivalent and the objective refraction spherical equivalent
8. Pupil size less than 2.5 mm in either eye prior to dilation at ambient light of 8-15 lux prior to the Baseline visit
9. A history of herpes (of any kind) in either eye
10. Cataract surgery and/or refractive surgery in either eye
11. Known contraindication, hypersensitivity and/or allergy to any study drugs or excipients
12. Any acute illness (e.g. acute infection) within 48 hours of first study drug administration, which is considered of significance by the Investigator
13. Participation in another clinical trial with drugs received within 30 days of Screening
14. Pregnant or currently lactating women

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with ≥ 2 lines improvement from Baseline in best distance corrected near visual acuity (monocular and binocular) | Baseline to end of treatment (up to 3 days)

SECONDARY OUTCOMES:
Change from Baseline in uncorrected near visual acuity (monocular and binocular) | Baseline to end of treatment (up to 3 days)
Change from Baseline in best corrected distance visual acuity (monocular and binocular) | Baseline to end of treatment (up to 3 days)
Change from Baseline in pupil diameter and appearance | Baseline to end of treatment (up to 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Klienman, Prof., Principal Investigator — Director, Cataract Service, Ophthalmology Department, Kaplan Medical Center, Rehovot, Israel; Zvi Segal, Dr., Principal Investigator — Director of Ophthalmology Department, Western Galilee Medical Center, Nahariya, Israel
Locations (2):
- Israel (2):
  - Ophthalmology Department, Western Galilee Medical Center, Nahariya
  - The Department of Ophthalmology, Kaplan Medical Center, Rehovot